CLINICAL TRIAL: NCT07297836
Title: Descriptionof Professional Practices Regarding Treatment of Non-vital Primary Teeth Among Dental Surgeons in France
Brief Title: Professional Practices Regarding Treatment of Non-vital Primary Teeth Among Dental Surgeons in France
Acronym: DTNV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9765
Record Dates: First submitted 2025-12-02; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pulpitis - Irreversible
Keywords: Pulpectomy; Pulp necrosis; Primary teeth; Non-vital primary teeth; Irreversible pulpitis; Natural exfoliation; Lesion Sterilization; Tissue Repair; Topical antibiotics; Pulpitis - Irreversible
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When faced with primary teeth affected by irreversible pulpitis or pulp necrosis, extraction is often the preferred option for practitioners, although validated alternatives exist, notably pulpectomy, which has high success rates when performed correctly. Recommended by the American Academy of Pediatric Dentistry, this technique relies on rigorous disinfection and the use of materials adapted to natural exfoliation. Low-stress treatment (LSTR), although more controversial due to the use of topical antibiotics, can also be considered in certain clinical situations. However, data on French practices in this area are very limited, hence the need to evaluate practitioners' treatment choices, their potential reservations, and the criteria guiding their decisions.

ELIGIBILITY:
Inclusion Criteria:

* Being a dentist treating children

Exclusion Criteria:

* Being a dentist treating children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dentist treating children
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Description of professional practices regarding the treatment of non-vital primary teeth by dentists in France | Up to 1 year
  There is no evaluation to be carried out in this study; It is just a matter of collecting and analyzing the professional practices of dental surgeons who treat children.
  The professional practices of dentists are collected through an anonymous questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine et Chirurgie Bucco-dentaires - CHU de Strasbourg - France, Strasbourg, France